CLINICAL TRIAL: NCT06968078
Title: Relationship Between Smartphone Addiction and Neck Angle and Balance in University Students
Brief Title: Smartphone Addiction in University Students
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-004
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smartphone addict: It will consist of individuals identified as addicted according to the smartphone addiction scale.
- Normal: It will consist of individuals who are normally determined according to the smartphone addiction survey.

SUMMARY:
Smartphone usage has increased significantly in the last decade and smartphones have changed our lives to a great extent. Smartphone usage has advantages as well as disadvantages and therefore brings phone addiction with it. Smartphone addiction is defined as excessive use of smartphones to the extent that it disturbs the daily lives of users. It has been stated in the literature that phone addiction can cause some disorders in individuals. Changes in neck posture and balance may be among the symptoms affected in this context. However, the relationship between excessive smartphone usage and neck proprioception, angle and balance is not clear in the literature. Therefore, the aim of our study was to examine the relationship between smartphone addiction and neck angle, proprioception and balance.

DETAILED DESCRIPTION:
Smartphones are not only a source of communication, information and entertainment today, but are also used for taking photos, playing games and surfing the internet. For this reason, smartphone use is increasing. In addition to all these advantages, excessive use of smartphones also brings phone addiction. Smartphone addiction is defined as the excessive use of smartphones to the extent that they disturb the daily lives of users. Smartphone addiction causes various disorders in individuals for this reason. The most important of these disorders are neck pain, anxiety and visual fatigue. In addition, excessive phone use can cause problems in neck movements and change neck posture. Therefore, sensory functions can also be affected. However, when the literature is examined, the relationship between smartphone use and neck proprioception, angle and balance is unknown. Therefore, this study aims to examine the relationship between smartphone addiction and neck angle, proprioception and balance and to compare these parameters according to smartphone addiction.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45
* Having a smartphone
* Volunteer to participate in the study

Exclusion Criteria:

* Individuals reporting orthopaedic, neurological, psychiatric and otological diseases will not be included in the study.
* Also, individuals with diagnosed vertigo will not be included in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who use smartphones and do not have any chronic diseases will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-04 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Smartphone addiction scale | Baseline
  It will be evaluated with The Smartphone Addiction Scale. The scale consists of 33 questions and is scored between 33-198. The higher the score, the higher the addiction.
Neck posture | Baseline
  Neck posture will be evaluated using neck angle. The craniocervical angle of individuals will be evaluated using a photographic method.
Neck proprioception | Baseline
  It will be evaluated with CROM. The deviation angle from 30 degrees will be recorded for flexion, extension, right and left lateral flexion and rotation. As the deviation angle increases, proprioception worsens.
Body balance | Baseline
  Balance will be assessed with static posturography. With static posturography, participants will be subjected to open and closed eyes on hard and soft surfaces. In this way, the static balance skills of the participants will be determined.
Dizziness imbalance | Baseline
  It will be evaluated with the Vertigo Dizziness Imbalanca-Symptom Scale. The scale consists of 14 items and is scored between 0-70. Lower scores indicate high symptom frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Gunes, Study Director — Karabuk University; Emre Söylemez, PhD, Principal Investigator — Karabuk University; Aydın Sinan Apaydın, PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhazmi AA, Alzahrani SH, Baig M, Salawati EM, Alkatheri A. Prevalence and factors associated with smartphone addiction among medical students at King Abdulaziz University, Jeddah. Pak J Med Sci. 2018 Jul-Aug;34(4):984-988. doi: 10.12669/pjms.344.15294. PMID 30190766
- [Background] Kumar VA, Chandrasekaran V, Brahadeeswari H. Prevalence of smartphone addiction and its effects on sleep quality: A cross-sectional study among medical students. Ind Psychiatry J. 2019 Jan-Jun;28(1):82-85. doi: 10.4103/ipj.ipj_56_19. Epub 2019 Dec 11. PMID 31879452